CLINICAL TRIAL: NCT03181152
Title: The Application of Impulse Oscillometry on the Differential Diagnosis of ACOS,Asthma and COPD.
Brief Title: The Application of Impulse Oscillometry on the Diagnosis of ACOS,Asthma and COPD.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YIZHUO GAO, master, Shengjing Hospital
Other Study IDs: SJHX-002
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Asthma-COPD Overlap Syndrome; Asthma; COPD; Diagnoses Disease
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ACOS group: Impulse Oscillometry Bronchial Dilation Test if needed
  Interventions: Diagnostic Test: Impulse Oscillometry
- Asthma group: Impulse Oscillometry Bronchial Dilation Test if needed
  Interventions: Diagnostic Test: Impulse Oscillometry
- COPD group: Impulse Oscillometry Bronchial Dilation Test if needed
  Interventions: Diagnostic Test: Impulse Oscillometry

INTERVENTIONS:
Diagnostic Test: Impulse Oscillometry — 1，Before the experiment, the patient is arranged to rest 10min. 2, IOS: The patient take seats, body relax, make sure the mouthpiece is fully covered by mouth, then clip nose with both hands to cover both sides of the cheek, and then calm breathing 1 minutes, the computer is automatically collected data calculation and print out the measurement results.
  3, Bronchial Dilation Test: The patient is asked to take IOS again after gaven aerosol inhalation of 200g salbutamol for 15min, the computer is automatically collects the data computation and prints the measurement result.
  Other Names: Bronchial Dilation Test

SUMMARY:
To Assess the Utility of Impulse Oscillometry on a Differential Diagnosis among the Patients with ACOS,asthma and COPD over Age 40.

DETAILED DESCRIPTION:
ACOS,asthma and COPD are prevalent diseases with similar manifestations and different type airway impairments. The differential diagnosis is not easy because the patients always complain of the similar symptoms and are not able to complete spirometry well.

Impulse Oscillometry System (IOS) is capable of identifying airway obstruction and reactions to bronchodilators by providing impedance data and curves. IOS is also a patient-friendly and valuable tool with minimal demands on patient and requiring only passive cooperation.

IOS is a tool to measure lung function during tidal breathing. The output is a measure of respiratory impedance (Zrs), which include the respiratory resistance (Rrs) and respiratory reactance (Xrs) measured over a range of frequencies (usually from 3 to 35 Hz).

The main objective of this study is to investigate the ability of IOS to measure small airway disease by providing different impedance profiles for participants with ACOS,asthma and COPD. Another objective of this study is to investigate the differential ability to identify three diseases by measuring airway impedance and reactions to bronchodilators.

First,participants completed the IOS test.Second,participants inhaled salbutamol for 200g 15 minutes to repeat the IOS.The investigators collect these 2 data for analysis.

ELIGIBILITY:
Inclusion Criteria:

- 1.1 ACOS:

1. Patient is older than 40 years old.
2. There are characteristics of bronchial asthma and COPD.
3. There is a history of exposure to risk factors.
4. Existence of persistent airflow limitation: After the application of bronchodilators, FEV1/FVC<0.7, and lung function proved reversible exhalation.
5. The existence of reversible airflow limitation: Bronchial Dilation Test positive.

1.2Asthma: 1)Patient is older than 40 years old. 2)History of reversible respiratory symptoms. 3) non-smokers. 4)lung function:At least one time proved that the airflow limitation: Bronchial Dilation Test positive.

5)previously diagnosed asthma. 1.3COPD:

1. Patient is older than 40 years old.
2. Complaints about dyspnea, chronic cough or expectoration.
3. There is a history of exposure to risk factors.
4. Existence of persistent airflow limitation: After the application of bronchodilators, FEV1/FVC<0.7.
5. The existence of irreversible airflow limitation: Bronchial Dilation Test negative.

Exclusion Criteria:

- 2.1 Combining other respiratory diseases that affect airflow,such as lung cancer, tuberculosis, pneumonia and bronchiectasis.

2.2 At the time doing lung function test, the factors that affect the airflow limitation are not stopped or just stopped with the time interval not long enough to meet the test standard.

2.3 Using special accompanying medication. For example, patients with drugs such as glucocorticoid.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients that meet one of the diganosis:ACOS,Asthma and COPD.
  2. Without factors in exclusion criteria.
  3. Over 40 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Data:physiological parameter of IOS in ACOS/Asthma/COPD group | 2018-8-30
  Parameter :
  parameter about respiratory impedance (Zrs): Z5,Zrs; parameter about respiratory resistance (Rrs)：R5,R20,R10,R35,R5%,R20%,R10%;R35%,△R5-R20,△R10-R20,△R5-R10； parameter about respiratory reactance (Xrs): X5,X20,X35, other parameter: fres,△AX, Alx,
Primary Data:physiological graph of IOS in ACOS/Asthma/COPD group | 2018-8-30
  Graph:Z-Time graph, impedance-volume graph,impedance-spectrum graph, structural parameter graph, Intrabreath graph.
Primary Data:physiological parameter of IOS combing BDT(Bronchial Dilation Test) in ACOS/Asthma/COPD group | 2018-8-30
  Parameter (IOS combing BDT):
  parameter about respiratory impedance (Zrs): Z5,Zrs; parameter about respiratory resistance (Rrs)：R5,R20,R10,R35,R5%,R20%,R10%;R35%,△R5-R20,△R10-R20,△R5-R10； parameter about respiratory reactance (Xrs): X5,X20,X35, other parameter: fres,△AX, Alx,
Primary Data:physiological graph of IOS combing BDT(Bronchial Dilation Test) in ACOS/Asthma/COPD group | 2018-8-30
  Graph(IOS combing BDT):Z-Time graph, impedance-volume graph,impedance-spectrum graph, structural parameter graph, Intrabreath graph.

CONTACTS AND LOCATIONS:
Overall Officials: LI ZHAO, Doctor, Study Director — SHENJING HOSPTIAL Affiliated to CHINA MEDICAL UNIVERSITY
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No